CLINICAL TRIAL: NCT01312610
Title: Effect of Chronic Orange Juice Consumption on Cognitive Function in Healthy Older Adults
Brief Title: Orange Juice Consumption and Cognitive Function
Acronym: OJOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor Jeremy Spencer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: UReading_2010_OJOC
Record Dates: First submitted 2011-03-09; First posted 2011-03-10 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Nerve Degeneration
Keywords: orange juice; cognitive function; flavonoids; flavanones
MeSH Terms: conditions — Nerve Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High flavonone orange juice drink (Experimental)
  Interventions: Dietary Supplement: High flavanone orange juice
- Control orange juice drink (Placebo Comparator): Juice drink matched for sugar content
  Interventions: Dietary Supplement: Control orange juice

INTERVENTIONS:
Dietary Supplement: High flavanone orange juice — High flavonone orange juice drink.
  Other Names: Frozen Orange Juice; Department of Citrus, Florida, USA.
  Arms: High flavonone orange juice drink
Dietary Supplement: Control orange juice — Orange beverage, low flavanone content, matched for total carbohydrate content, individual sugar profile, vitamin C
  Arms: Control orange juice drink

SUMMARY:
This study is investigating the effect of 8 weeks of orange juice supplementation on executive function in healthy older adults. The study is a controled, double-blind, crossover trial and involves a 8 week supplementation with a high flavonone orange juice and a carbohydrate-matched control. Volunteers consume 500ml of either the test juice or the control juice per day for an 8 week period. There is then an 8 week washout period before subjects proceed to the other arm of the study. Subjects are randomly assigned to either arm at the beginning of the study. Measures of cognitive function will be administered pre and post both test and control interventions. Blood pressure will also be measured and blood and urine samples will be collected to assess absorption of from the juice. A sub-sample of volunteers will undergo MRI imaging pre- and post intervention to acquire cerebral blow flow information.

ELIGIBILITY:
Inclusion Criteria:

* In good general health i.e. no major health condition such as diabetes
* BMI < 30
* Cholesterol < 6 and BP < 150/90
* Not on blood pressure medication or blood thinning medication such as aspirin - No learning difficulty such as dyslexia

Exclusion Criteria:

* Diabetes
* Gastro-intestinal disease
* High BMI
* Cholesterol and BP
* Smoker
* On blood pressure medication or blood thinning medication such as aspirin
* Dyslexic/dyspraxic
* Depression or history of depression

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Executive function - Attention | change in attention from baseline and 8 weeks
  Assessment by human cognitive test battery delivered by computer and human operator. Assessments will be carried out at baseline and at the end of each intervention arm.

SECONDARY OUTCOMES:
Plasma flavanones | change from baseline to 8 weeks
  By High performance liquid chromatography
Blood pressure | change from baseline to 8 weeks
  Blood pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, PhD, Principal Investigator — University of Reading; Laurie T. Butler, PhD, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Kean RJ, Lamport DJ, Dodd GF, Freeman JE, Williams CM, Ellis JA, Butler LT, Spencer JP. Chronic consumption of flavanone-rich orange juice is associated with cognitive benefits: an 8-wk, randomized, double-blind, placebo-controlled trial in healthy older adults. Am J Clin Nutr. 2015 Mar;101(3):506-14. doi: 10.3945/ajcn.114.088518. Epub 2015 Jan 14. PMID 25733635